CLINICAL TRIAL: NCT01647243
Title: Effect of Preoperative Strength Training on Postoperative Quadriceps Strength and Ability of Function in Patients With Total Knee Arthroplasty in Fast Track Regi
Brief Title: Preoperative Strength Training in Patients With Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M-20110181
Record Dates: First submitted 2012-07-13; First posted 2012-07-23 (Estimated); Last update posted 2012-07-23 (Estimated); Status verified 2012-07

CONDITIONS: Osteoarthritis, Knee
Keywords: Knee osteoarthritis; Total knee arthroplasty; Preoperative training; Strength training
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Preoperative strength training (Experimental): Progressive strength training on group basis four weeks before the operation and progressive strength training on group basis four weeks after the operation
  Interventions: Other: Preoperative strength training
- Living as usual (No Intervention): The patients are living as usual the last 4 weeks before operation

INTERVENTIONS:
Other: Preoperative strength training — Progressive strength training on group basis (not more than 3 subjects) 3 sessions weekly starting 4 weeks before the operation, in total 12 sessions Strength training 3 sessions weekly 4 weeks postsurgery
  Other Names: Strength training; Preoperative training
  Arms: Preoperative strength training

SUMMARY:
The purpose of this study is to investigate if preoperative strength training will result in faster recovery and higher level of function six weeks after total knee arthroplasty (TKA).

DETAILED DESCRIPTION:
Reduced strength of the quadriceps muscle is a common clinical finding in patients with Knee Osteoarthritis and this seems to play a central role in the development of the disease. The strength of the quadriceps muscle have been shown to be reduced by 20-40% as compared to age-matched healthy controls and this decrease in muscle strength have been closely associated with a reduced level of function and increase of pain. Furthermore, it has been demonstrated that the preoperative strength of the quadriceps muscle in patients undergoing TKA, is associated with the level of function one year after surgery. Compared to the level before the operation, an additional operation-induced reduction of the strength of the quadriceps muscle up to 60% as has been demonstrated. Presumably, an optimizing of the strength of the quadriceps muscle could counteract the impact of the expected postoperative loss of muscle strength to such an extent that the loss will be of less clinical significance. It is hypothesized that an optimizing of the strength of the quadriceps muscle may have a favorable effect on the postoperative rehabilitation program and shorten the period of convalescence.

ELIGIBILITY:
Inclusion Criteria:

* Planned TKA at the Aarhus University Hospital or Region Hospital Silkeborg,
* Living in Aarhus Municipality,
* Primary knee osteoarthritis or secondary osteoarthritis after meniscectomy or ligament injury

Exclusion Criteria:

* Unstable blood pressure,
* Neuromuscular or neurodegenerative disease,
* Comprehension or dementia problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-10 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Primary outcome: Sit-to-stand test | Change from Baseline 6 weeks preoperative in Sit-to-Stand at 6 weeks postoperative
  Ability of function test

SECONDARY OUTCOMES:
Isokinetic: Quadriceps 60 gr./sek | 6 weeks and 1 week before the operation, 1 week, 6 weeks, 12 weeks and 1 year after the operation
  Muscle strength test in dynamometer
Isokinetic: Hamstrings 60 gr./sek | 6 weeks and 1 week before the operation, 1 week, 6 weeks 12 weeks and 1 year after the operation
  Muscle strength test in dynamometer
Isometric: Quadriceps (70 gr. flexion) | 6 weeks and 1 week before the operation and 11 week, 6 weeks, 12 weeks and 1 year after the operation
  Muscle strength test in dynamometer
Isometric: Hamstrings (20 gr. flexion) | 6 weeks and 1 week before the operation, 1 week, 6 weeks, 12 weeks and 1 year after the operation
  Muscle strength test in dynamometer
Rate of force development (flexion and extension) | 6 weeks and 1 week before the operation, 1 week, 6 weeks, 12 weeks and 1 year after the operation
  Muscle test in dynamometer
Timed Up and Go | 6 weeks and 1 week before the operation, 1 week, 6 weeks, 12 weeks and 1 year after the operation
  Ability of function test
10 meter walk test | 6 weeks and 1 week before the operation, 1 week, 6 weeks, 12 weeks and 1 year after the operation
  Ability of function test
6 minute walk test | 6 weeks and 1 week before operation, 1 week, 6 weeks, 12 weeks and 1 year after the operation
  Ability of function test
Knee injury and Osteoarthritis Outcome Score (KOOS) | 6 weeks and 1 week before operation, 1 week, 6 weeks, 12 weeks and 1 year after the operation
  Disease-specific questionnaire
Oxford Knee Score (OKS) | 6 weeks before the operation and 6 weeks after
  Disease-specific questionnaire
EuroQol-5 dimensions (EQ-5D) | 6 weeks and 1 week before the operation, 1 week, 6 weeks, 12 weeks and 1 year after the operation
  Generic questionnaire for self-rated health
Short-Form Health Survey (SF 12) | 6 weeks before the operation and 1 year after
  Generic questionnaire for self-rated health
Background data questionnaire | 6 weeks and 1 week before the operation, 1 week, 6 weeks, 12 weeks and 1 year after the operation
  Questionnaire about pain, medicine use, alcohol intake, smoking, education, job
Range of motion of the knee | 6 weeks and 1 week before the operation, 1 week, 6 weeks, 12 weeks and 1 year after the operation
  Extension of the knee Flexion of the knee
Body mass index | 6 weeks and 1 week before the operation, 1 week, 6 weeks, 12 weeks and 1 year after the operation
  Weight/height2

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Soeballe, Professor, Study Chair — Aarhus University Hospital, Department of orthopaedic, Tage Hansensgade 2, 8000 Aarhus C
Locations (1):
- Aarhus University hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Skoffer B, Dalgas U, Maribo T, Soballe K, Mechlenburg I. No Exacerbation of Knee Joint Pain and Effusion Following Preoperative Progressive Resistance Training in Patients Scheduled for Total Knee Arthroplasty: Secondary Analyses From a Randomized Controlled Trial. PM R. 2018 Jul;10(7):687-692. doi: 10.1016/j.pmrj.2017.11.002. Epub 2017 Nov 9. PMID 29129608
- [Derived] Skoffer B, Maribo T, Mechlenburg I, Hansen PM, Soballe K, Dalgas U. Efficacy of Preoperative Progressive Resistance Training on Postoperative Outcomes in Patients Undergoing Total Knee Arthroplasty. Arthritis Care Res (Hoboken). 2016 Sep;68(9):1239-51. doi: 10.1002/acr.22825. Epub 2016 Jul 28. PMID 26713665